CLINICAL TRIAL: NCT00972556
Title: Comparison of Mineral Trioxide Aggregate and 20% Formocresol in Pulpotomized Human Primary Molars :A Long-Term Follow-Up Study
Brief Title: Comparison of Mineral Trioxide Aggregate (MTA) and 20% Formocresol (FC) in Pulpotomized Human Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Department of Dentistry, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200905028R
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Dental Caries; Pulpitis
Keywords: Mineral Trioxide Aggregate; Formocresol; pulpotomy; primary molar; treatment outcome
MeSH Terms: conditions — Dental Caries; Pulpitis | interventions — ProRoot MTA; formocresol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GMTA (Experimental)
  Interventions: Drug: Gray Mineral Trioxide Aggregate (GMTA)
- 20% FC (Active Comparator)
  Interventions: Drug: Diluted (20%) Formocresol (DFC)

INTERVENTIONS:
Drug: Gray Mineral Trioxide Aggregate (GMTA) — Once hemorrhage from the pulp chamber is under control using direct pressure of a sterile cotton pellet, pulp stumps are covered with a MTA paste, obtained by mixing 0.2g GMTA powder with sterile water in a powder to liquid ratio of 3:1 in weight. The GMTA will be then immediately covered with a zinc-oxide eugenol base (IRM) material.
  Other Names: ProRoot MTA
  Arms: GMTA
Drug: Diluted (20%) Formocresol (DFC) — After the pulp hemostasis is achieved with direct pressure of a sterile cotton pellet, a sterile cotton pellet dampened with 20% DFC will be placed in contact with the pulp for 5 minutes, followed by the immediate placement of a zinc-oxide eugenol base (IRM) material.
  Other Names: Buckley's Formo Cresol
  Arms: 20% FC

SUMMARY:
This prospective clinical randomized controlled trial is established to compare the clinical, radiographic, and histological treatment outcomes between MTA and FC in pulpotomized human primary molars at 6, 12, 18, 24 month post-treatment and to test the hypothesis that Gray Mineral Trioxide Aggregate (GMTA) is a viable alternative to Diluted (20%) Formocresol (DFC) in pulpotomies treatment of human primary molars.

DETAILED DESCRIPTION:
1. Background: Formocresol (FC) is the most widely used pulpotomy medicament in the primary dentition. There are concerns associated with this medicament, primarily the carcinogenicity of the chemical and internal resorption of the treated tooth. Recently, Mineral Trioxide Aggregate (MTA) has been suggested with preliminary studies showing promising results.
2. Study design: This is a prospective clinical randomized controlled trial (RCT), which will be performed at Department of Dentistry, National Taiwan University Hospital, to compare the treatment outcomes between MTA and FC in pulpotomized human primary molars and to evaluate whether GMTA is a viable alternative to DFC in pulpotomies treatment of human primary molars.
3. Hypotheses:

   * Null Hypotheses: there is no clinical, radiographic, or histological difference between GMTA and DFC at 6, 12, 18, 24 month post-treatment when used as a pulp dressing agent in pulpotomized primary molars.
   * Alternative Hypotheses: There is a statistically significant difference between GMTA and DFC as a pulpotomy agent. GMTA shows clinical and/or radiographic and/or histological success as a dressing material following pulpotomy in primary human molars and may be a suitable replacement for DFC in primary molar pulpotomy.
4. Specific Aims:

   * The primary aims of this investigation are:

     1. Compare the clinical and radiographic results of GMTA with DFC pulpotomies on vital human primary molars at 6, 12, 18, and 24 months post-operatively.
     2. Assess intraradicular histological changes of the pulpal tissue and root dentin following pulpotomy treatment with GMTA or DFC.
   * The secondary aims of this investigation are:

     1. Assess the outcome of GMTA by multiple operators that have been calibrated to the methods of mixing and placing the material.
     2. Assess whether sex, tooth type, arch, and age of patient at time of treatment influence the overall success rate of GMTA pulpotomies.
     3. Compare the radiographic success of the two materials based on both the traditional radiographic assessment criteria adopted by the American Academy of Pediatric Dentistry (AAPD) and the alternative radiographic success criteria adopted by Zurn et al. 2000.
     4. To serve as a basis for future research in the comparison of GMTA and DFC pulpotomies. This will include larger sample size, longer follow-up periods, and a collaborative study with UM group (Prof. Jan C. Hu).

ELIGIBILITY:
Inclusion Criteria:

* Primary first or second molars with normal pulp, reversible, or irreversible pulpitis, that have vital carious pulp exposures due to caries and whose pulp bled upon entering the pulp chamber.
* Teeth in which hemostasis could be achieved with pressure of a saline dampened sterile cotton pellet prior to medicament/material placement.
* No clinical symptoms or evidence of pulp degeneration, such as excessive bleeding from the root canal, history of swelling, mobility, or sinus tracts.
* Patients with percussion sensitivity or spontaneous and persistent pain but where hemostasis could be achieved with pressure of sterile cotton pellet.
* No radiographic signs of internal or external root resorption, inter-radicular and/or periapical bone destruction, or furcation radiolucency.
* No more than one-third physiologic root resorption has occurred.
* Teeth had not previously been pulpally treated.
* Teeth deemed to be restorable with posterior stainless steel crowns.

Exclusion Criteria:

* Not present

Ages: 30 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
clinically and radiographically outcomes | 6, 12, 18, and 24 months

SECONDARY OUTCOMES:
histological outcome | when the subjective tooth physically exfoliates from oral cavity

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Ling Lee, PhD, Principal Investigator — Department of Dentistry, National Taiwan University Hospital; Hsiao-Hua Chang, MS, Study Chair — Department of Dentistry, National Taiwan University Hospital
Locations (1):
- Department of Dentistry, National Taiwan University Hospital, Taipei, Taiwan